CLINICAL TRIAL: NCT01332825
Title: cAMP Levels in the Nose
Brief Title: cAMP (Cyclic Adenosine Monophosphate) Levels in the Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Greg Davis, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 39352-A
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Olfactory Disorder
Keywords: olfaction; smell dysfunction
MeSH Terms: conditions — Anosmia; Olfaction Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- olfactory dysfunction (No Intervention): subjects diagnosed with olfactory dysfunction
- normal olfaction, no saline (No Intervention): no smell dysfunction, not randomized to saline nasal irrigation for 7 days
- normal olfaction (Other): normal olfaction, randomized to saline nasal irrigation for 7 days
  Interventions: Other: saline nasal irrigation

INTERVENTIONS:
Other: saline nasal irrigation — subjects irrigate with nasal saline daily for one week
  Arms: normal olfaction

SUMMARY:
The purpose of this study is to determine the normal distribution of nasal tissue cathelicidin antimicrobial peptides (cAMP) levels in subjects with normal smell and subjects with smell dysfunction. The investigators will also look at the effect of nasal saline irrigation on olfaction and cAMP levels and if nasal irrigation is capable of harvesting olfactory cilia. The investigators hypothesize that nasal saline will have no effect on olfaction and will be inadequate to harvest olfactory cilia.

DETAILED DESCRIPTION:
The investigators will recruit 40 subjects: 10 with olfactory dysfunction and 30 with normal olfaction. The normal olfaction group will be randomized (15-15)to either daily saline nasal irrigation for one week or no irrigation. Normal olfaction subjects will be seen for two visits, olfactory dysfunction for one. All subjects will complete an UPSIT (smell identification test)and a co-morbidity form. All subjects will have a brief nasal exam and then have nasal cells collected by means of a curette on one side and a cytobrush on the other. All subjects will receive Afrin and lidocaine, to improve visualization and for comfort during cell collection. Subjects will then complete a Comfort Scale related to the methods of cell collection. Normal olfaction subjects randomized to nasal irrigation will receive instructions on how to do it and the irrigation results will be collected for analysis along with the nasal cells. At their return visit, normal olfaction subjects will repeat the UPSIT and the comfort scale--all normal olfaction subjects will have a repeat cell collection. Subjects randomized to nasal irrigation will also complete a transition scale which asks if they feel the irrigation made a difference in their sense of smell. Subjects are compensated for time with a gift card.

ELIGIBILITY:
Inclusion Criteria:

Normal olfactory function cohort:

* self-reported normal smell function
* age greater than 18 years

Olfactory dysfunction cohort:

* ICD9 diagnostic code for olfactory dysfunction
* idiopathic olfactory dysfunction
* age greater than 18 years

Exclusion Criteria:

* allergy to lidocaine
* active upper respiratory infection
* previous nasal or sinus surgery
* current tobacco use
* unable to give consent due to language barrier, cognitive or medical issues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
UPSIT | 7 days
  validated, scratch and sniff smell identification test

CONTACTS AND LOCATIONS:
Overall Officials: Greg E Davis, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States